CLINICAL TRIAL: NCT02003482
Title: Prospective Observational Trial of Serial CT Imaging for Evaluation of Dosimetric/Volumetric Changes During IMRT for Head/Neck Cancer
Brief Title: Prospective Trial of Serial CT Imaging for Evaluation of Dosimetric/Volumetric Changes During IMRT for Head/Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Cristiane Takita, MD, Professor of Clinical, University of Miami
Other Study IDs: 20060212
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Intensity modulated radiation therapy; IMRT; Anatomic Changes; Postoperative; Unresectable
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postop IMRT for Head/Neck cancer: CT for Radiation Treatment Planning
  Interventions: Radiation: Postop IMRT for head/neck cancer; Device: CT for Radiation Treatment Planning
- Chemo/IMRT for bulky Head/Neck cancer: CT for Radiation Treatment Planning
  Interventions: Radiation: Postop IMRT for head/neck cancer; Device: CT for Radiation Treatment Planning

INTERVENTIONS:
Radiation: Postop IMRT for head/neck cancer — Patients will be enrolled in study through the duration of their radiation therapy, approximately 6-8 weeks. After which time no further evaluations will be made.
  Other Names: IMRT
Device: CT for Radiation Treatment Planning — Treatment planning CT scans will be required to define tumor, clinical, and planning target volumes. This study requires CT scans prior to initiation of treatment then again on the third and sixth week of radiation treatment
  Other Names: CT Simulation

SUMMARY:
Anatomical changes that take place during Intensity modulated radiation therapy (IMRT) treatments for cancers of the head and neck cause significant dosimetric changes.

DETAILED DESCRIPTION:
The investigator's hypothesis is that those patients with bulky head and neck cancers who undergo definitive radiation therapy with or without chemotherapy have changes in their dose distribution that lead to significant changes in dose to tumor and/or normal tissue. It is possible for these dosimetric changes could occur in either those patients who undergo resection or not. In this study those patients who have undergone a resection will be stratified separately for analysis, however, this study is not powered to detect a difference between the two groups. The rational for stratification into an operated group of patients is that these patients will also lose weight in treatment and will provide us a detection of the magnitude of change in dose caused by weight loss independent of tumor shrinkage.

ELIGIBILITY:
Inclusion Criteria:

* AJCC pathological stage I-IV cancers of the head and neck meeting the following criteria:

  * If gross total resection is performed it must be completed within 7 weeks of registration
* Site of tumor origin in the nasopharynx, oral cavity, oropharynx, parotid, larynx, or hypopharynx (excluding lip, or sinuses)
* Pretreatment evaluations required for eligibility include:

  * History and physical examination within four weeks prior to study entry
  * Dental evaluation with management according to the guidelines in Appendix IV prior to start of radiation
  * Serum pregnancy test, if applicable, within one week prior to study entry; urine dipstick test on the first day of treatment
  * Radiographic Studies: Pre-operative CT or MRI of the primary tumor and neck for clinical staging is required
* Patients must be ≥ 18 years of age.
* Women of childbearing potential (WOCBP) must be willing to consent to using effective contraception while on treatment.
* Pregnant women are ineligible as radiation therapy involves unforeseeable risks to the embryo or fetus. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG], or in accordance with local regulations, whichever is more sensitive).
* Patients must sign a study-specific informed consent form prior to registration.

Exclusion Criteria:

* Histology positive for melanoma.
* Gross (visible or palpable) disease left after surgery.
* Less than gross total resection or patients requiring staged surgery.
* Prior head and neck radiotherapy.
* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologic stage I-IV cancers of the head and neck (site of tumor origin nasopharynx, parotid, oral cavity, oropharynx, larynx, or hypopharynx,) either following gross total resection and requiring postoperative XRT for high-risk features or undergoing definitive concurrent chemo-radiation.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2006-05-09 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Volumetric/Dosimetric Changes During IMRT for bulky and postoperative head/neck patients | 7 weeks
  To evaluate whether those patients undergoing standard intensity modulated radiation therapy (IMRT) for bulky and postoperative head and neck cancers demonstrate significant anatomic changes, causing dosimetric/volumetric changes during treatment which lead to under-dosing of tumor and/or over dosing of critical structures.

SECONDARY OUTCOMES:
Number of Participants Requiring Re-Planning During the Course of IMRT for bulky and postoperative Head and Neck Cancer | 7 weeks
  To determine whether patients undergoing standard IMRT for head and neck cancers require re-planning during the course of therapy, due to volumetric or dosimetric changes.
Length of Time Required for Replanning of Radiation Therapy | 7 weeks
  To estimate what the appropriate time course should be for re-planning of radiation therapy if it is deemed necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Takita, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States